CLINICAL TRIAL: NCT07107191
Title: The Relationship Between Dysfunctional Breathing and Physical Fitness in Older Adults: a Comparative Cross-sectional Study
Brief Title: Dysfunctional Breathing and Physical Fitness in Older Adults
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yunus Emre Tutuneken, Asst. Prof., Istinye University
Other Study IDs: 2025/203
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Dysfunctional Breathing; Older Adults
Keywords: physical fitness; dysfunctional breathing; older adults
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Data will be collected from all participants in assessmnet group.

SUMMARY:
The global aging trend will continue to challenge healthcare systems, making it increasingly important to preserve quality of life and independence among older adults. Physical fitness will remain a crucial factor for maintaining autonomy, yet aging will naturally lead to declines in respiratory function, muscle strength, balance, and flexibility. Dysfunctional breathing (DB), characterized by abnormal respiratory patterns without organic pathology, will become a growing public health concern in the elderly. Although symptoms such as breathlessness, fatigue, and anxiety will likely limit physical activity, the specific effects of DB on physical fitness in older adults will not yet be well understood. This study will aim to investigate the effects of DB on physical fitness components in older individuals and determine whether these effects are independent of demographic variables such as age and body mass index (BMI). The study will compare physical fitness levels between older adults with and without DB and will evaluate the predictive value of DB for physical performance outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Regularly monitored (followed) for at least six months
* Possess sufficient cognitive ability to communicate
* Able to perform activities of daily living independently or with minimal assistance
* No history of respiratory disease within the past three months
* No current acute illness

Exclusion Criteria:

* Advanced dementia or significant cognitive impairment
* A diagnosis of cardiopulmonary disease (e.g., COPD, congestive heart failure)
* A history of malignancy
* Serious musculoskeletal conditions
* Major surgery within the past six months
* Neurological or orthopedic problems that limit physical activity
* Refused to participate in the study
* Inability to complete the measurement procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: individuals aged sixty-five and older
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Nijmegen Questionnaire | 4 weeks
  The NQ evaluates and identifies respiratory dysfunction, unexplained respiratory symptoms, and HV syndrome symptoms. It contains 16 questions addressing neurological, cardiovascular, respiratory, gastrointestinal, and psychological factors. The questionnaire uses a 5-point Likert scale, with total scores ranging from 0 to 64. Higher scores suggest a greater likelihood of respiratory dysfunction and HV syndrome. A score above 23 indicates a possible DB diagnosis.
Senior Fitness Test Battery | 4 weeks
  To assess physical fitness levels, the Senior Fitness Test Battery , developed by Rikli and Jones, is administered, comprising six tests: chair sit-stand, weightlifting, chair sit-lie, 2-minute step, 8-step stand-walk, and back scratching.
30-Second Chair Stand Test | 4 weeks
  This test measures lower-body muscle strength. The participant sits in a 43.18 cm high chair with a straight back, feet flat on the floor, and arms crossed over the chest. Upon the "start" command, they stand up and sit down repeatedly as many times as possible within 30 seconds.
Arm Curl Test | 4 weeks
  This test assesses upper-body strength. The participant sits on the edge of a chair facing their dominant arm. They extend and flex their elbow for 30 seconds while holding a dumbbell (2.27 kg [5 lb] for women, 3.63 kg [8 lb] for men). Before testing, each participant was shown and explained the procedure, performing two or three practice attempts without weights. Once understood, the test commenced.
Two-Minute Step Test | 4 weeks
  This test is used to evaluate aerobic endurance. To perform the test, the distance from the anterior iliac crest to the midpoint of the patella was measured while the subject was standing straight.
Eight-Foot Up and Go Test | 4 weeks
  Eight-Foot Up and Go Test evaluates agility and dynamic balance. A person sitting upright in the center of a chair with their back resting against the backrest is asked to place both hands on their knees, keep their feet flat on the floor, and, upon the command "start," walk around a cone located 2.44 meters away and return to the chair as quickly as possible. The time taken (in seconds) to complete the test is recorded.
Chair Sit and Reach Test | 4 weeks
  Chair Sit and Reach Test measures lower-body flexibility. This modified sit-and-reach test uses a straight-backed chair with a seat height of 43.18 cm and a 46 cm ruler.
Back Scratch Test | 4 weeks
  This test evaluates upper extremity flexibility, especially shoulder flexibility. The subject stands, externally rotates one arm over their shoulder with the palm facing back and fingers extended, trying to reach the lowest point on their back.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunus Emre TÜTÜNEKEN, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided